CLINICAL TRIAL: NCT07077720
Title: COMPARISON OF THE EFFECT OF DISTAL ADDUCTOR CANAL BLOCK COMBINED WITH GENICULAR NERVE BLOCK OR PERIARTICULAR INJECTION ON POSTOPERATIVE QOR-15 IN TOTAL KNEE ARTHROPLASTIES: A RANDOMIZED CONTROLLED STUDY
Brief Title: COMPARISON OF THE EFFECT OF DISTAL ADDUCTOR CANAL BLOCK COMBINED WITH GENICULAR NERVE BLOCK OR PERIARTICULAR INJECTION ON POSTOPERATIVE QOR-15 IN TOTAL KNEE ARTHROPLASTIES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Muhammed Çağrı Sarıarslan, research assistant, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 29.01.2025-E.180706
Record Dates: First submitted 2025-07-01; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Pain; Recovery
Keywords: Total Knee Arthroplasty; Genicular nerve bloc; periarticular injection; QoR-15
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Spinal; Bupivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grup G (Active Comparator): Genicular nerve block
  Interventions: Procedure: genicular nerve block; Procedure: Addukctor canal block; Procedure: Spinal Anesthesia with Bupivacaine and Morphine
- Grup P (Active Comparator): Periarticular injecrion
  Interventions: Procedure: periarticular injection; Procedure: Addukctor canal block; Procedure: Spinal Anesthesia with Bupivacaine and Morphine

INTERVENTIONS:
Procedure: genicular nerve block — genicular nerve block with a total of 15 mL of 0.25% bupivacaine preoperatively
  Arms: Grup G
Procedure: periarticular injection — periarticular injection prepared by the surgical team containing 8 mg morphine, 40 mg methylprednisolone, 0.3 mg adrenaline, 750 mg cefazolin, and 110 mg bupivacaine.
  Arms: Grup P
Procedure: Addukctor canal block — Addukctor canal block with 15ml %0.25 bupivacaine
Procedure: Spinal Anesthesia with Bupivacaine and Morphine — Spinal Anesthesia with Bupivacaine(isobaris 15-18mg) and Morphine(100mcg)

SUMMARY:
Objective: This study compares the effects of genicular nerve block (GNB) and periarticular injection (PAI), added to distal adductor canal block (ACB), on postoperative recovery quality (QoR-15), morphine use, and pain scores after total knee arthroplasty (TKA).

Methods: Sixty patients received spinal anesthesia and distal ACB, then were randomized to GNB (Group G, n=30) or PAI (Group P, n=30). QoR-15, morphine consumption, VAS pain scores, nausea/vomiting, and side effects were evaluated.

DETAILED DESCRIPTION:
Objective: Total knee arthroplasty (TKA) is a common surgical procedure for knee pathologies of various etiologies, where postoperative pain management is critical for early mobilization and rehabilitation. Different blockade techniques targeting the femoral, obturator, and sciatic nerves, which provide sensory innervation to the knee, are evaluated in terms of analgesic efficacy and preservation of motor function. The adductor canal block (ACB) targets the saphenous nerve without affecting motor function, whereas periarticular injection (PAI) and genicular nerve block (GNB) provide more comprehensive analgesia by blocking other branches of the femoral nerve as well as the obturator and sciatic nerves. This study aims to compare the effects of GNB and PAI, applied in addition to distal ACB, on postoperative recovery quality measured by the Quality of Recovery-15 (QoR-15) score, morphine consumption, and pain scores in patients undergoing TKA.

Materials and Methods: This single-center, randomized, prospective study included patients over 18 years of age with ASA physical status I-III who were scheduled for total knee arthroplasty under spinal anesthesia. All patients received spinal anesthesia with 15 mg isobaric bupivacaine combined with 100 mcg intrathecal morphine. Additionally, all patients underwent ultrasound-guided distal adductor canal block. Patients were randomized into Group G (n=30) and Group P (n=30). Group G received preoperative genicular nerve block (5+5+5 ml of 0.25% bupivacaine), whereas Group P received intraoperative periarticular injection administered by the surgical team, consisting of 8 mg morphine, 40 mg methylprednisolone, 0.3 mg adrenaline, 750 mg cefazolin and 110 mg bupivacaine. The primary outcome measure was the quality of recovery evaluated by the Quality of Recovery-15 (QoR-15) questionnaire at 24 hours postoperatively. Secondary outcomes included morphine consumption at 2., 6., 12. and 24 hours postoperatively, resting and movement Visual Analog Scale (VAS) pain scores, postoperative nausea and vomiting (PONV) scores, and the incidence of adverse effects such as respiratory depression, urinary retention, and pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for knee arthroplasty
* Patients classified as ASA I, II, or III
* Patients aged 18 years and older

Exclusion Criteria:

* Patients with a known allergy to any of the drugs used in the study
* Presence of infection near the puncture site
* History or presence of neurological disorders (e.g., transient ischemic attack, syncope, dementia, etc.)
* Known coagulation disorders
* History of alcohol or substance abuse
* Impaired consciousness
* Chronic opioid use equal to or exceeding 60 mg of oral morphine equivalents per day
* Pre-existing neuropathic pain
* Hepatic failure, renal failure, or cardiac insufficiency
* Uncontrolled diabetes mellitus
* Pregnant or breastfeeding women
* Refusal or inability to provide written informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Postoperative 24th hour qor-15 | Postoperative 24th hour
  Postoperative 24th hour qor-15 score

SECONDARY OUTCOMES:
Postoperative 2nd, 6th, 12th, and 24th hour morphine consumption | Postoperative 2nd, 6th, 12th, and 24th hour
  Postoperative 2nd, 6th, 12th, and 24th hour morphine consumption
Postoperative 2nd, 6th, 12th, and 24th hour resting VAS score | Postoperative 2nd, 6th, 12th, and 24th hour
  Postoperative 2nd, 6th, 12th, and 24th hour resting VAS score
Postoperative 2nd, 6th, 12th, and 24th hour movement VAS score | Postoperative 2nd, 6th, 12th, and 24th hour
  Postoperative 2nd, 6th, 12th, and 24th hour movement VAS score
Postoperative 2nd, 6th, 12th, and 24th hour adverse effects | Postoperative 2nd, 6th, 12th, and 24th hour
  Postoperative 2nd, 6th, 12th, and 24th hour adverse effects

CONTACTS AND LOCATIONS:
Locations (1):
- Bezmialem vakıf üniversitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No